CLINICAL TRIAL: NCT06914336
Title: Hepatic Doppler to Assess Venous Congestion During Invasive Mechanical Ventilation
Brief Title: Hepatic Doppler to Assess Venous Congestion During Invasive Mechanical Ventilation (DOHECOV)
Acronym: DOHECOV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC25.0048 - DOHECOV
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Congestion, Venous
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to investigate venous congestion using hepatic vein doppler for ICU patients with invasive mechanical ventilastion. The primary outcome is the systolic to diastolic hepatic vein velocity ratio S/D . The objective is to find a significant association between S/D and different congestion indicators.

ELIGIBILITY:
Inclusion Criteria:

* intubated for more than 24 hours

Exclusion Criteria:

* Chronic end-stage renal disease on admission
* Atrial Fibrillation
* Cirrhosis
* Portal thrombosis
* Refusal to participate
* non-opposition could not be obtained from themselves or their trusted support person in the event of incapacity
* Under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were included if they were intubated for more than 24 hours. Patients were excluded if they had chronic end-stage renal disease on admission, atrial fibrillation, cirrhosis, portal thrombosisrefusal to participate, whose non-opposition could not be obtained from themselves or their trusted support person in the event of incapacity or if they were under legal protection.
  S/D velocity ratio was measured as well as veinous congesion parameters such as weight variation, cumulative fluid balance, peripheral edema, central venous pressure, urine output and acute kidney failure KDIGO stage.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Systolic to diastolic hepatic vein velocity ratio S/D | 24 hours after intubation and after every 48 hours until extubation up to 12 weeks
  Relate S/D ratio to clinical data on venous congestion: input/output balance, weight variation, renal insufficiency, diuresis, edema.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement